CLINICAL TRIAL: NCT05016726
Title: Intravascular Lithotripsy and/or Mechanical Debulking Multicenter Registry for the Treatment of Complex Calcified Coronary Arteries: the ROLLING-STONE.
Brief Title: Intravascular Lithotripsy and/or Mechanical Debulking for Severely Calcified Coronary Artery Lesions
Acronym: ROLLING-STONE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SS Annunziata Hospital, Savigliano (Other)
Responsible Party: Principal Investigator, Marco Pavani, MD, SS Annunziata Hospital, Savigliano
Other Study IDs: 001
Record Dates: First submitted 2021-07-14; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Atherectomy, Coronary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Intravascular Lithotripsy — Intravascular Lithotripsy and/or Rotational Atherectomy and/or Orbital Atherectomy to the target vessel prior to placing a coronary stent.
  Other Names: Rotational Atherectomy; Orbital Atherectomy

SUMMARY:
To evaluate intra-procedural and long-term effects of intravascular lithotripsy with the ShockWave System and/or non-balloon mechanical debulking devices, prior and/or after coronary stenting in an angiographically well-defined group of patients with complex calcified coronary artery lesions.

DETAILED DESCRIPTION:
At present age, there are few real-world data published about the use of intravascular lithotripsy. Its safety and possible procedural complications remain unclear, and the effects of combination with other plaque-modification devices are unknown. Finally, there are few data about long-term outcomes in the real-life setting.

Subject Population: Subjects ≥ 18 years of age with de novo, calcified coronary artery lesions presenting with Stable CAD or Acute Coronary Syndromes, that are suitable for percutaneous coronary intervention (PCI). Approximately 400 subjects at 20 sites will be enrolled. Subjects will be followed through discharge, 30 days, 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. ≥18 years of age;
2. Native coronary artery disease suitable for PCI;
3. Patients with stable ischemic heart disease or unstable ischemic heart disease (Unstable Angina, Non-ST Elevation Myocardial Infarction, ST-Elevation Myocardial Infarction), patients with concomitant cardiogenic shock.
4. Patient or legally authorized representative, signs a written Informed Consent form to participate in the study, prior to any study-mandated procedures;

Angiographic Inclusion Criteria:

1. The target vessel reference diameter must be ≥2.5 mm.
2. De novo coronary lesions or calcific in-stent restenosis or suboptimal stent expansion in a severely calcified coronary segment: Unprotected or Protected Left Main, LAD, LCfx, Ramus, RCA.
3. Angiographic stenosis > 70% or stenosis > 50% and < 70% with FFR < 0.80 or iFR < 0.90 or IVUS or OCT minimum lumen area ≤4.0 mm²;
4. Evidence of calcification at the lesion site: angiographic calcifications (Mintz el al Classification) are described as : None/mild, Moderate (radio-opacities noted only during cardiac cycle prior to contrast injection) severe calcification: radio-opacities seen without cardiac motion prior to contrast injection, usually affecting both sides of the arterial lumen.

Exclusion Criteria:

1. Patient is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint;
2. Patient is pregnant or nursing (a negative pregnancy test is required for women of child-bearing potential within 7 days prior to enrollment);
3. Patient has an allergy to imaging contrast media which cannot be adequately pre-medicated;
4. Patient has an active systemic infection on the day of the index procedure with either fever, leukocytosis or requiring intravenous antibiotics;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a novel diagnosis of complex severe calcified coronary artery confirmed by core-lab analysis of coronary angiograms or other intravascular imaging available
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Freedom from major adverse cardiac events (MACE) within 30 days of the index procedure. | within 30 days of index procedure
  The primary safety endpoint was freedom from major adverse cardiac events (MACE) within 30 days of the index procedure.
  Definition of MACE:
  Composite of
  * cardiac death;
  * myocardial infarction (MI): CK-MB level >3 times the upper limit of lab normal (ULN) value with or without new pathologic Q waves at discharge (periprocedural MI) and using the Fourth Universal Definition of Myocardial Infarction beyond discharge (spontaneous MI)
  * target vessel revascularization: revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure.
Number of Participants With Procedural Success | within 30 days of index procedure
  The primary effectiveness endpoint was procedural success defined as stent delivery with a residual stenosis <20% (Image Core Laboratory-Assessed) and without intra-procedural MACE.

SECONDARY OUTCOMES:
Residual stenosis < 30% | intra-procedural
  Stent delivery with ≤30% residual stenosis and without serious angiographic complications.
Serious angiographic complications | intra-procedural
  Severe dissection (Type D to F), perforation, abrupt closure, persistent slow flow or persistent no reflow, pericardial effusion, access-site complications (in-hospital).
MACE at 6 and 12 months | at 6 and 12 months
  Cardiac death, myocardial infarction (MI), or target vessel revascularization (TVR).
Target lesion failure (TLF) | at 30 days, 6 and 12 months.
  Cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or ischemia-driven target lesion revascularization (ID-TLR) by percutaneous or surgical methods at 30 days, 6 and 12 months.
Other clinical secondary outcomes | at 30 days, 6 months nd 12 months.
  All death, cardiac death, MI, target vessel MI (TV-MI), ischemia-driven TVR (ID-TVR), ID-TLR, ID-non-TLR, ID-non-TVR, all revascularizations (ID and non-ID), and stent thrombosis (ARC definite, probable, definite or probable)
Intraprocedural secondary outcome | intra-procedure
  1.Minimal Lumen Diameter pre-stenting and post-stenting (mm at QCA evaluation)
Intraprocedural secondary outcome | intra-procedure
  Minimal Lumen Area (mm2) pre-stenting and post stenting (IVUS/OCT)
Intraprocedural secondary outcome | intra-procedure
  QFR value at the end of the procedure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cerrato E, Pavani M, Zecchino S, Leoncini M, Zanda G, Abdirashid M, Cordone S, Nicolino A, Franze A, Bernardi A, Lio V, Boi A, Marengo G, Presutti DG, Vadala P, Secco GG, Conrotto F, Vergallo R, Menozzi A, Berchialla P, Tomassini F, Patti G, Musumeci G, Chinaglia A, Varbella F. Intravascular Lithotripsy or Mechanical Debulking in Complex Calcified Coronary Arteries: Multicenter, Prospective ROLLING STONE Study. JACC Cardiovasc Interv. 2026 Jan 24:S1936-8798(25)03190-5. doi: 10.1016/j.jcin.2025.11.033. Online ahead of print. PMID 41609534